CLINICAL TRIAL: NCT03695172
Title: Comparison of TAP, Anterior QL, or ESP Block for Elective Cesarean Section
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Decline of eligible participants
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100742
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Pain, Postoperative; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of three treatment groups, TAP, QL, or ESP blocks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- TAP block (Active Comparator): Patients will receive bilateral TAP blocks after delivery and within one hour of skin closure with 25 mL of 0.2% ropivacaine with epinephrine 1:400,000 per side.
  Interventions: Drug: Ropivacaine; Procedure: TAP block
- QL block (Active Comparator): Patients will receive bilateral QL blocks after delivery and within one hour of skin closure with 25 mL of 0.2% ropivacaine with epinephrine 1:400,000 per side.
  Interventions: Drug: Ropivacaine; Biological: QL block
- ESP block (Active Comparator): Patients will receive bilateral ESP blocks after delivery and within one hour of skin closure with 25 mL of 0.2% ropivacaine with epinephrine 1:400,000 per side.
  Interventions: Drug: Ropivacaine; Procedure: ESP block

INTERVENTIONS:
Drug: Ropivacaine — Patients will be randomly assigned to receive one three blocks (TAP, QL, ESP)after delivery of baby with ropivicaine
Procedure: TAP block — Patient will receive bilateral TAP blocks after delivery and within one hour of skin closure with 25 mL of 0.2% ropivacaine with epinephrine 1:400,000 per side.
  Arms: TAP block
Biological: QL block — Patients will receive bilateral QL blocks after delivery and within one hour of skin closure with 25 mL of 0.2% ropivacaine with epinephrine 1:400,000 per side.
  Arms: QL block
Procedure: ESP block — Patients will receive bilateral ESP blocks after delivery and within one hour of skin closure with 25 mL of 0.2% of ropivacaine with epinephrine 1:400,000 per side.
  Arms: ESP block

SUMMARY:
The purpose of this prospective single center, randomized study is to determine if ultrasound guided Transversus Abdominis Plane (TAP), Quadratus Lumborum (QL), and Erector Spinae Plane (ESP) blocks decrease opioid consumption in subjects undergoing elective cesarean section.

DETAILED DESCRIPTION:
The typical anesthetic for cesarean section at Duke University Hospital includes a spinal or combined spinal epidural anesthetic with intrathecal dosing of 1.4-1.6 mL bupivacaine HCl 0.75%, 15 mcg fentanyl, and 150 mcg morphine. If the epidural component of a combined spinal epidural anesthetic is used, the subject will be withdrawn from the study. Patients also receive rectal acetaminophen 975 mg prior to incision; intravenous (IV) ondansetron 4 mg, IV metoclopramide 10 mg, IV famotidine 20 mg and IV dexamethasone 4 mg intraoperatively; and IV ketorolac 15 mg prior to skin closure. There will be no change to this typical practice.

Patients who consent to be in this study will be randomized to receive one of three truncal nerve blocks using an online randomization program by the study PI (AK/EG): (1) ultrasound-guided bilateral classic TAP block; (2) ultrasound-guided bilateral anterior QL (also known as transmuscular or QL type 3) block; (3) ultrasound-guided bilateral ESP block at the level of T9. These nerve blocks will be performed after delivery and within one hour of skin closure with 25 mL of 0.2% ropivacaine with epinephrine 1:400,000 per side. Nerve blocks will be performed by a dedicated and trained group of regional anesthesiologists. This non-blinded regional anesthesiologist will save an ultrasound image after local anesthetic administration while the needle is still in position on each side. The study team will review these images to ensure a high quality of block performance.

Patients will have standard postoperative pain medication orders, including acetaminophen 975 mg PO Q6H for 4 days (scheduled, starting 6 hours after intraoperative rectal dose), ketorolac 15 mg IV Q6H for 24 hours (scheduled, starting 6 hours after intraoperative dose), ibuprofen 600 mg PO Q6H for 3 days (scheduled, starting 24 hours after first dose of ketorolac) and oxycodone 5-10mg PO Q3-4H PRN for 4 days. If patients are unable to tolerate oral medication or oxycodone is insufficient, rescue medications may be ordered: IV morphine 1-2 mg or IV hydromorphone 0.3-0.5 mg Q4H as needed. There is no change from the standard postoperative order sets used for patients after cesarean section.

Subjects' verbal pain scores at rest and with movement as well as opioid consumption will be recorded at 2, 6, 24, and 48 hours postoperatively. Additionally, the amount of antiemetics and antipruritics used will also be recorded at the above time points. These scores will be entered into a Duke University Hospital REDCap database. Subjects will also be sent a survey assessing their satisfaction with pain control one week after discharge via email or telephone. This information will be collected via Duke University Hospital REDCap.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Physical Status 1-3
2. Age greater than or equal to 18 years
3. Scheduled for elective cesarean section
4. English speaking

Exclusion Criteria:

1. ASA Physical Status 4-5
2. Diagnosis of chronic pain
3. Chronic opioid use (opioid use in the past 3 months)
4. Preoperative use of SSRIs (Celexa, Lexapro, Prozac, Paxil), SNRIs (Cymbalta, Effexor), gabapentin, or pregabalin (Lyrica)
5. Inability to cooperate with or understand protocol
6. Inability to communicate pain scores or need for analgesia
7. Infection at the site of block placement
8. Intolerance or allergy to local anesthetics
9. Neurologic deficit or disorder
10. Blood thinning disorder or taking anticoagulant medication
11. BMI > 50 kg/m2
12. Suspected or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
13. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance
14. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Kumar, MD, Principal Investigator — Duke
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcus MA, Brodner G. Are opioids contraindicated as postoperative pain relief for patients who are breast-feeding their newborn? Curr Opin Anaesthesiol. 2001 Jun;14(3):287-9. doi: 10.1097/00001503-200106000-00001. No abstract available. PMID 17019104
- [Background] Marcus H, Gerbershagen HJ, Peelen LM, Aduckathil S, Kappen TH, Kalkman CJ, Meissner W, Stamer UM. Quality of pain treatment after caesarean section: Results of a multicentre cohort study. Eur J Pain. 2015 Aug;19(7):929-39. doi: 10.1002/ejp.619. Epub 2014 Nov 21. PMID 25413847
- [Background] Bateman BT, Cole NM, Maeda A, Burns SM, Houle TT, Huybrechts KF, Clancy CR, Hopp SB, Ecker JL, Ende H, Grewe K, Raposo Corradini B, Schoenfeld RE, Sankar K, Day LJ, Harris L, Booth JL, Flood P, Bauer ME, Tsen LC, Landau R, Leffert LR. Patterns of Opioid Prescription and Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):29-35. doi: 10.1097/AOG.0000000000002093. PMID 28594763
- [Background] Osmundson SS, Schornack LA, Grasch JL, Zuckerwise LC, Young JL, Richardson MG. Postdischarge Opioid Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):36-41. doi: 10.1097/AOG.0000000000002095. PMID 28594766
- [Background] Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. Am J Obstet Gynecol. 2016 Sep;215(3):353.e1-353.e18. doi: 10.1016/j.ajog.2016.03.016. Epub 2016 Mar 17. PMID 26996986
- [Background] Eslamian L, Jalili Z, Jamal A, Marsoosi V, Movafegh A. Transversus abdominis plane block reduces postoperative pain intensity and analgesic consumption in elective cesarean delivery under general anesthesia. J Anesth. 2012 Jun;26(3):334-8. doi: 10.1007/s00540-012-1336-3. Epub 2012 Feb 22. PMID 22354671
- [Background] Fusco P, Scimia P, Paladini G, Fiorenzi M, Petrucci E, Pozone T, Vacca F, Behr A, Micaglio M, Danelli G, Cofini V, Necozione S, Carta G, Petrini F, Marinangeli F. Transversus abdominis plane block for analgesia after Cesarean delivery. A systematic review. Minerva Anestesiol. 2015 Feb;81(2):195-204. Epub 2014 Apr 16. PMID 24739207
- [Background] Factor D, Chin KJ. Transversus abdominis plane block in lower segment cesarean section: a question of block failure or lack of efficacy? Reg Anesth Pain Med. 2010 Jul-Aug;35(4):404-5. doi: 10.1097/AAP.0b013e3181e66f01. No abstract available. PMID 20588155
- [Background] Loane H, Preston R, Douglas MJ, Massey S, Papsdorf M, Tyler J. A randomized controlled trial comparing intrathecal morphine with transversus abdominis plane block for post-cesarean delivery analgesia. Int J Obstet Anesth. 2012 Apr;21(2):112-8. doi: 10.1016/j.ijoa.2012.02.005. Epub 2012 Mar 10. PMID 22410586
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Kadam VR. Ultrasound guided quadratus lumborum block or posterior transversus abdominis plane block catheter infusion as a postoperative analgesic technique for abdominal surgery. J Anaesthesiol Clin Pharmacol. 2015 Jan-Mar;31(1):130-1. doi: 10.4103/0970-9185.150575. No abstract available. PMID 25788791
- [Background] Kadam VR, Howell S. Ultrasound-guided continuous transmuscular quadratus lumborum block- L4 or L2 level catheter insertion for analgesia in open abdominal surgery: Case series. Indian J Anaesth. 2018 Jul;62(7):555-557. doi: 10.4103/ija.IJA_242_18. No abstract available. PMID 30078860
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Luis-Navarro JC, Seda-Guzman M, Luis-Moreno C, Chin KJ. Erector spinae plane block in abdominal surgery: Case series. Indian J Anaesth. 2018 Jul;62(7):549-554. doi: 10.4103/ija.IJA_57_18. PMID 30078859
- [Background] Tulgar S, Selvi O, Kapakli MS. Erector Spinae Plane Block for Different Laparoscopic Abdominal Surgeries: Case Series. Case Rep Anesthesiol. 2018 Feb 18;2018:3947281. doi: 10.1155/2018/3947281. eCollection 2018. PMID 29670771
- [Background] Yamak Altinpulluk E, Garcia Simon D, Fajardo-Perez M. Erector spinae plane block for analgesia after lower segment caesarean section: Case report. Rev Esp Anestesiol Reanim (Engl Ed). 2018 May;65(5):284-286. doi: 10.1016/j.redar.2017.11.006. Epub 2018 Jan 17. English, Spanish. PMID 29352577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Block | QL Block | ESP Block
Started | 5 | 4 | 3
Completed | 4 | 3 | 3
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block | QL Block | ESP Block | Total
Number analyzed (Participants) | 4 | 3 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 3 | 10
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 34.25 [26 to 39] | 28 [25 to 32] | 31.33 [27 to 39] | 32 [25 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 2 | 1 | 5
  White | 1 | 1 | 2 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Consumption
Description: Amount of opioid in milligrams.
Time Frame: 2 hours postoperatively
Measure: Mean (Full Range); unit: mg
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
mg | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Postoperative Opioid Consumption
Description: Amount of opioid
Time Frame: 6 hours postoperatively
Measure: Mean (Full Range); unit: mg
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
mg | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Primary Outcome: Postoperative Opioid Consumption
Description: Amount of opioid
Time Frame: 24 hours postoperatively
Measure: Mean (Full Range); unit: mg
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
mg | 0 [0 to 0] | 11.66 [0 to 20] | 0 [0 to 0]

4. Primary Outcome: Postoperative Opioid Consumption
Description: Amount of opioid
Time Frame: 48 hours postoperatively
Measure: Mean (Full Range); unit: mg
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
mg | 0 [0 to 0] | 38.3 [0 to 70] | 15 [0 to 25]

5. Primary Outcome: Postoperative Pain Scores
Description: Visual Analog Scale at rest with 0 being no pain and 10 being the worst pain imaginable
Time Frame: 2 hours postoperatively
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
units on a scale | .25 [0 to 1] | 0 [0 to 0] | .33 [0 to 1]

6. Primary Outcome: Postoperative Pain Scores
Description: Visual Analog Scale at rest with 0 being no pain and 10 being the worst pain imaginable
Time Frame: 6 hours postoperatively
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
units on a scale | .25 [0 to 1] | 0 [0 to 0] | 1 [0 to 2]

7. Primary Outcome: Postoperative Pain Scores
Description: Visual Analog Scale at rest with 0 being no pain and 10 being the worst pain imaginable
Time Frame: 24 hours postoperatively
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
units on a scale | .75 [0 to 1] | 2 [0 to 3] | 1 [0 to 2]

8. Primary Outcome: Postoperative Pain Scores
Description: Visual Analog Scale at rest with 0 being no pain and 10 being the worst pain imaginable
Time Frame: 48 hours postoperatively
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
units on a scale | 1.3 [0 to 2] | 1.6 [0 to 3] | 3 [0 to 5]

9. Secondary Outcome: Number of Participants Requiring Antipruritics
Time Frame: 2 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Requiring Antipruritics
Time Frame: 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Requiring Antipruritics
Time Frame: 24 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 0 | 3 | 0

12. Secondary Outcome: Number of Participants Requiring Antipruritics
Time Frame: 48 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 0 | 2 | 0

13. Secondary Outcome: Number of Participants Requiring Antiemetics
Time Frame: 2 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 2 | 1 | 1

14. Secondary Outcome: Number of Participants Requiring Antiemetics
Time Frame: 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 2 | 0 | 2

15. Secondary Outcome: Number of Participants Requiring Antiemetics
Time Frame: 24 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 2 | 1 | 2

16. Secondary Outcome: Number of Participants Requiring Antiemetics
Time Frame: 48 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 4 | 3 | 3
Participants | 2 | 1 | 1

17. Secondary Outcome: Overall Satisfaction With Pain Control
Description: Satisfaction Rating, with 0 being not at all satisfied and 10 being completely satisfied
Time Frame: 1 week postoperatively
Population: Date not collected.
Arm/Group | TAP Block | QL Block | ESP Block
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | TAP Block | QL Block | ESP Block
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03695172/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT03695172/ICF_001.pdf